CLINICAL TRIAL: NCT03207490
Title: sEMG Based-Rehabilitation of Hand and Fingers After Stroke
Brief Title: Robotics for Rehabilitation of Hand and Fingers After Stroke
Acronym: sERF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Camillo, Venezia, Italy (Other)
Responsible Party: Principal Investigator, Andrea Turolla, Laboratory Head, IRCCS San Camillo, Venezia, Italy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Prot. 2014.14
Record Dates: First submitted 2016-01-12; First posted 2017-07-02 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Stroke
Keywords: Hand; Rehabilitation; sEMG
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Intervention is provided by a robotic device for hand motion, controlled by closed loop surface electromyography (sEMG)
Oversight: Data Monitoring Committee: No

ARMS (1):
- Robot group (Experimental): Receive 1 hour of AMADEO (robot-assisted therapy) for the hand and 1 hour of daily standard rehabilitation therapy
  Interventions: Device: AMADEO

INTERVENTIONS:
Device: AMADEO — Robot therapy: 1-Degrees-Of-Freedom (1DOFs) robot training for flexion and extention movements of the hand.
  Standard rehabilitation therapy includes speech, physical, occupational therapies and group activities
  Other Names: Robot-assisted therapy for the hand

SUMMARY:
The major issue for a person who has suffered a stroke is the severe impairment affecting the hand and the high risk to have a poor recovery associated. Innovative approaches are needed in the next future, translating recent advances from neuro-engineering, into feasible devices for rehabilitation care. The FP7-EU project MYOSENS aims to translate known motor control logic from sEMG prosthetic control, to rehabilitation robotics. The target is to promote the closing of sensory-motor loop on the basis of intention to move, as detected from residual sEMG (i.e. Extensor Digitorum Communis, Flexor Digitorum Profundus).

DETAILED DESCRIPTION:
The objectives of this pilot study are:

* to assess whether a clinical and kinematic effect might be induced providing a closed-loop control by sEMG signal for robot (i.e. Amadeo ®) assisted therapy of hand function
* to determine safety and feasibility of including robotic therapy into daily rehabilitation programs after stroke.

A total of 20 patients has been recruited, all of them received on daily basis 1 hour of robot therapy in adjunction to 1 hour of standard therapy. Overall the hour of robotic therapy include both subject preparation (15 minutes to place surface electrodes on the forearm and set the right position of sitting and upper limb) and delivery of exercises. The treatment protocol includes passive and active training of flexion and extension movements of the fingers. The passive part lasts 5 minutes, while the active one provides 25 total minutes divided into 5 exercises. The robot therapy lasts 15 consecutive sessions, 5 times a week, for 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from first stroke, ischemic and/or hemorrhagic
* Score between 1 and 3 at the upper-limb sub-item of the Italian version of the National Institute of Health Stroke Scale, IT-NIHSS (Pezzella et al. 2009)
* Score lower than 100 out of a total of 126 at the Functional Independence Measure (FIM) scale.
* Less than 45 cubes carried in one minute whit the affected hand at the Box and Bocks Test.

Exclusion Criteria:

* Non-stabilized fractures
* Diagnosis of depression
* Traumatic brain Injury
* Untreated or drug resistant seizures.
* Severe ideomotor apraxia
* Severe neglect
* Patients participating in other rehabilitation treatments for the upper-limb (e.g. virtual reality treatment, motor imagery).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-07; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change at Box and Block Test (BBT) | Before treatment, then 3 weeks after
  Hand dexterity is measured by means of the BBT. The patient has to carry as much cubes as possible, one by one, from a container to another one in one minute. The test is performed with both hands.

SECONDARY OUTCOMES:
Change at Functional Independence Measure scale (FIM) | Before treatment, then 3 weeks after
  FIM is an 18-item scale that assesses the degree of autonomy in carrying out activities of daily living (total score = 126 points).
Change at Reaching Performance Scale (RPS) | Before treatment, then 3 weeks after
  RPS assesses the ability of subjects to reach an object (a cone). The cone is placed at both 4-cm (close) and 30-cm (far) distance from the subject. The subject is asked to reach and grab the cone if possible. The observer evaluates the quality of reaching instead of the grip strength (Total score = 36 points).
Change at Modified Ashworth Scale (MAS) | Before treatment, then 3 weeks after
  Spasticity is measured using the MAS of five muscles: Pectoralis major, biceps, wrist flexors, flexor digitorum superficialis, flexor digitorum profundus (Total score = 20 points).
Change at Nine Hole Pegboard Test (NHPT) | Before treatment, then 3 weeks after
  NHPT measures the dexterity of the hand. Patient should insert 9 pins in the board. There are 9 pins. The number of pins inserted in 50 sec are registered or if the patient inserted 9 pins, then the time is registered.
Change at Fugl-Meyer Assessment Scale: Upper Extremity Motor Function (F-M UE) | Before treatment, then 3 weeks after
  Motor function of the upper limb is measured by means of the Fugl-Meyer Scale. There are 3 values: 0 (severe impairment), 1 (moderate impairiment), 2 (preserved function)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Turolla, PhD, Principal Investigator — IRCCS San Camillo, Venezia, Italy
Locations (2):
- Tyromotion GmbH, Graz, Austria
- IRCCS San Camillo Hospital Foundation, Venice, Italy

REFERENCES:
- [Background] Hwang CH, Seong JW, Son DS. Individual finger synchronized robot-assisted hand rehabilitation in subacute to chronic stroke: a prospective randomized clinical trial of efficacy. Clin Rehabil. 2012 Aug;26(8):696-704. doi: 10.1177/0269215511431473. Epub 2012 Jan 19. PMID 22261813
- [Background] Sale P, Lombardi V, Franceschini M. Hand robotics rehabilitation: feasibility and preliminary results of a robotic treatment in patients with hemiparesis. Stroke Res Treat. 2012;2012:820931. doi: 10.1155/2012/820931. Epub 2012 Dec 26. PMID 23320252
- [Background] Stein J, Bishop L, Gillen G, Helbok R. Robot-assisted exercise for hand weakness after stroke: a pilot study. Am J Phys Med Rehabil. 2011 Nov;90(11):887-94. doi: 10.1097/PHM.0b013e3182328623. PMID 21952215
- [Background] Takahashi CD, Der-Yeghiaian L, Le V, Motiwala RR, Cramer SC. Robot-based hand motor therapy after stroke. Brain. 2008 Feb;131(Pt 2):425-37. doi: 10.1093/brain/awm311. Epub 2007 Dec 20. PMID 18156154